CLINICAL TRIAL: NCT03900182
Title: The Role of Hyperbaric Oxygen and Neuropsychological Therapy in Cognitive Function Following Traumatic Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 pandemic, patients can not receive hyperbaric oxygen therapy.
Sponsor: Hung-Chen Wang (Other)
Responsible Party: Sponsor-Investigator, Hung-Chen Wang, Attending physician; Associate professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201801854A3
Record Dates: First submitted 2019-03-25; First posted 2019-04-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Brain Injuries, Traumatic; Neuropsychology
Keywords: Traumatic brain injury; hyperbaric oxygen therapy; neuropsychological treatment; cognitive function; biomarkers.
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: After signing an informed consent form, the patients were invited for baseline evaluation. Included patients were randomized into two groups. The neuropsychological functions were the primary endpoints of the study. Secondary end point included quality of life evaluation. Evaluations were made by medical and neuropsychological practitioners who were blinded to patients' inclusion in the control-crossed or the treated groups.
  Patients in the treated group were evaluated three - at baseline, after 6 weeks of HBOT and after 6 weeks of neuropsychological treatment or no treatment. Patients in the crossover group were evaluated three times: baseline, after 6 weeks control period of no treatment, and after subsequent 6 weeks of HBOT. The post-HBOT neuropsycological evaluations were performed more than 1 week (1-2 weeks) after the end of the HBOT protocol. The following HBOT protocol was practiced: 30 daily sessions, 5 days/week, 60 minutes each, 100% oxygen at 1.5ATA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBO treated group (Active Comparator): Patients in the treated group were evaluated three - at baseline, after 6 weeks of HBOT and after 6 weeks of neuropsychological treatment or no treatment.
  Interventions: Device: Hyperbaric Oxygen Therapy
- crossover group (Sham Comparator): Patients in the crossover group were evaluated three times: baseline, after 6 weeks control period of no treatment, and after subsequent 6 weeks of HBOT
  Interventions: Device: Hyperbaric Oxygen Therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — The Hyperbaric Oxygen Therapy (HBOT) patients were placed in a chamber that was pressurized with air to 2.5 ATA during 15 min and were supplied 100% oxygen for 25 mins, followed by a 5-min air break. This cycle was repeated once and followed by 100% oxygen for 10 min, after which time the chamber was depressurized to 1 ATA over 15 min with 100% oxygen for a total treatment time of 100 min.
  Other Names: Neuropsychological Therapy

SUMMARY:
Traumatic brain injury (TBI) caused by accidents is a very important public health problem in Taiwan. There are many people with brain damage and cognitive dysfunction caused by traumatic brain injury every year. Currently, there is no effective treatment for cognitive dysfunction caused by traumatic brain injury. Evidence from clinical studies in recent years suggests that hyperbaric oxygen therapy may be a treatment for repairing nerves after brain injury.

Many studies have shown that oxidative stress and inflammatory responses play an important role in the pathogenesis of the central nervous system. In recent years, our research team has shown that oxidative stress and inflammatory response are significantly associated with the prognosis of patients with traumatic brain injury, cerebral hemorrhage, and stroke patients. More and more evidences also show that oxidative stress and inflammatory response play an important role in the neuropathological changes of mental cognitive sequelae after traumatic brain injury. This injury may be gradual from the time of head trauma. This process begins with the generation of oxidative stress and free radicals. When the cell repair and free radical scavenging system can not effectively overcome the excessive production of free radicals, an oxidative damage reaction will occur, causing a series of inflammatory cells and cytokines to be activated. Studies have also shown that when inhibiting those free radicals that produce oxidative stress, the neurological function and cognitive function of the head after trauma can be significantly improved.

It is becoming widely acknowledged that the combined action of hyperoxia and hyperbaric pressure leads to significant improvement in tissue oxygenation while targeting both oxygenand pressure-sensitive genes, resulting in improved mitochondrial metabolism with anti-apoptotic and anti-inflammatory effects. The investigators published an article this year showing that hyperbaric oxygen therapy can improve the prognosis of patients with acute stroke and increase endothelial progenitor cells in the systemic circulation.

The investigators plan to conduct this research project through hyperbaric oxygen therapy and neuropsychological therapy, and using scientific tests and neurocognitive function assessments. The investigators hope to answer the following questions: (1) Whether the treatment of hyperbaric oxygen can improve oxidative stress and inflammatory response after brain injury, and observe changes in biomarker concentration; (2) Whether hyperbaric oxygen therapy and neuropsychological therapy can improve cognitive function after brain injury; and (3) which biomarkers are factors that influence cognitive function prognosis.

DETAILED DESCRIPTION:
Research Methodology A prospective cohort study will be conducted. The follow-up periods are 18 weeks.

Diagnostic criteria of mild and moderate traumatic brain injury. Diagnostic criteria of traumatic brain injury will be according to (1) American Association of Neurosurgical Surgeons (AANS) Guidelines for The Management of Severe Head Injury; (2) YOUMANS Neurological Surgery Fifth Edition Guidelines for Traumatic Brain Injury.

Definitions and classifications Traumatic brain injury is defined as damage to the brain resulting from external mechanical force, such as rapid acceleration or deceleration, impact, blast waves, or penetration by a projectile. Consequently to the injury, brain function is temporarily or permanently impaired and structural damage may or may not be detectable with current imaging technology. TBI is usually classified based on severity, anatomical features of the injury, and the cause of the injury. The severity is assessed according to the loss of consciousness (LOC) duration, the post-traumatic amnesia (PTA), and the Glasgow coma scale (GCS) grading of the level of consciousness. Approximately (70-90%) of the TBI in the US are classified as mild TBI (mTBI) or concussion - LOC duration of 0-30 minutes, PTA duration of less than a day and GCS grade of 13-15. Post concussion syndrome (PCS) is a set of symptoms succeeding mTBI in most patients. The PCS symptoms include headache, dizziness, neuropsychiatric symptoms, and cognitive impairments. In most patients, PCS may continue for weeks or months, and up to 25% of the patients may experience prolonged PCS (PPCS) in which the symptoms last for over six months. Such individuals are at high risk for emotional and cognitive dysfunction, culminating in inability to carry out ordinary daily activities, work responsibilities and standard social relationships.

Hypotheses and Purpose:

In this study, the investigators hypothesize that the hyperbaric oxygen therapy in neurotherapeutics, in light of recent persuasive evidence for hyperbaric oxygen therapy efficacy in brain repair and of new understanding of brain energy management and response to damage. The investigators discuss the optimal timing of treatment, optimal dose-response curve (oxygenpressure levels), suitable candidates and promising future directions. The investigators speculate that these changes of biomarkers correlated with the hyperbaric oxygen therapy efficacy and the progression of neuropsychological testing during the 18 weeks follow-up.

The investigators plan to conduct this research project through hyperbaric oxygen therapy and neuropsychological therapy and using scientific tests and neurocognitive function assessments. The scientific tests including flow cytometry to evaluate the fraction of circulating activated platelets, the proportion of leukocytosis apoptosis, Erythrocyte assay of antioxidant enzymes and Enzyme-Linked Immunosorbent Assay (ELISA) for inflammatory markers.

Purpose:

1. To evaluate that whether the treatment of hyperbaric oxygen can improve oxidative stress and inflammatory response after brain injury, and observe changes in biomarker concentration.
2. To evaluate that whether hyperbaric oxygen therapy and neuropsychological therapy can improve cognitive function after brain injury.
3. To evaluate that which biomarkers are factors that influence the prognosis of cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury, mild and moderated.
* Age between 18 and 65 years old

Exclusion Criteria:

1. Penetrating injury, including gunshot injury
2. Combined with other major trauma which had unstable hemodynamics
3. Major systemic disease, such ESRD, liver cirrhosis, CHF, or a malignant disease
4. Evidence for alcoholism or any other addictive disorders, or known affective or other psychiatric disease or use of sedatives or neuroleptic medication
5. Known neurological disorders potentially affecting the central nervous system or severe recent life events that might have interfered with neuropsychological testing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Neuropsychological testing- Wechsler Adult Intelligence scale-III (WAIS-III) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  Subtests included the followings: Information with a measure of general knowledge, digit Span, vocabulary ability to define 35 words, arithmetic, comprehension, similarities, picture completion, picture arrangement, block design, digit symbol, and object assembly. The scores could further subscore into verbal comprehension, perceptual reasoning and working memory index.
Neuropsychological testing- Cognitive Ability Screening Instrument (CASI) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  includes tests of nine domains of cognitive function (attention, concentration, orientation, short and long-term memory, language ability, visual construction, word list generation, abstraction, and judgment), and the score ranges from 0 (worst) to 100 (best score).
Neuropsychological testing- mini-mental state examination (MMSE) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  The Mini-Mental State Examination (MMSE) test is a 30-point questionnaire. Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.
Neuropsychological testing- Short Form 36 questionnaire | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  The SF-36 taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scoring the SF-36 is a two-step process. First, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores.
Neuropsychological testing- The World Health Organization Quality of Life questionnaire (WHOQOL-BREF) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  questionnaire is a 26-item questionnaire that evaluates 4 domains of quality of life (QoL), namely Physical, Psychological, Social Relationships and Environment
Neuropsychological testing- Beck Depression Inventory | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used here differ from the original as such: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; and 29-63: severe depression.

SECONDARY OUTCOMES:
oxidative damage markers: Erythrocyte superoxide dismutase (SOD) activity | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  by a commercially available kit (Ransod, Randox Lab., Grumlin, UK) based on the method developed by McCord and Fridovich. The SOD activity is then measured by the degree of inhibition of this reaction. The assay will be carried out on washed red blood cells, by diluting the samples to give between 30 and 60% inhibition. Together with the kit, a standard is supplied, which is diluted to provide a range of standards and a calibration curve. A standard curve will be produced by plotting % inhibition for each standard against Log 10. The result will be multiplied by the appropriate dilution factor (100) and expressed in units/litre (U/L) of whole blood.
oxidative damage markers: Erythrocyte glutathione peroxidase (GPx) activity | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  Erythrocyte GPx activity will be measured using a commercially available kit (Ransel; Randox Lab, Crumlin, U.K.). The result obtained will be expressed in U/L of haemolysate and will be multiplied by the appropriate dilution factor to obtain the result in U/L of whole blood.
oxidative damage markers: serum malondialdehyde (MDA) content | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  Serum MDA will be measured using the thiobarbituric acid reactive substances (TBARS) assay. TBARS reagent (1 ml) will be added to a 0.5 ml aliquot of serum and heated for 20 minutes at 100°C. The antioxidant, butylated hydroxytoluene, will be added before heating the samples. After cooling on ice, samples will be centrifuged at 840 g for 15 mins and absorbance of the supernatant will be read at 532 nm. Blanks for each sample will be prepared and assessed in the same way to correct for the contribution of A532 to the sample. TBARS results will be expressed as MDA equivalents using 1,1,3,3-tetraethoxypropane.
oxidative damage markers: serum free thiol content | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  Plasma free thiols will be determined by directly reacting thiols with 5,5-dithiobis 2-nitrobenzoic acid (DTNB) to form 5-thio-2- nitrobenzoic acid (TNB). The amount of thiols in the sample will be calculated from the absorbance determined using extinction coefficient of TNB (A412 = 13,600 M-1cm-1).
Cytokines (IL-1β) by Enzyme-linked immunosorbent assays | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
Cytokines (IL-6) by Enzyme-linked immunosorbent assays | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
Cytokines (IL-10) by Enzyme-linked immunosorbent assays | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
Cytokines (TNF-α) by Enzyme-linked immunosorbent assays | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
endothelium-leukocyte activation (ICAM-1) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
endothelium-leukocyte activation ( VCAM-1) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
endothelium-leukocyte activation (E-selectin) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
endothelium-leukocyte activation (L-selectin) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  will be assayed in serum samples and quantified with a commercially available colorimetric ELISA.
neural inflammation markers (S-100) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  by Enzyme-linked immunosorbent assays; The values of intra- and inter-assay coefficients were around 5%. Concentration is expressed as pg/ml
neural inflammation markers (tau protein) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  by Enzyme-linked immunosorbent assays; The values of intra- and inter-assay coefficients were around 5%. Concentration is expressed as pg/ml
neural inflammation markers (MMP-2) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  by Enzyme-linked immunosorbent assays; The values of intra- and inter-assay coefficients were around 5%. Concentration is expressed as ng/ml
neural inflammation markers (MMP-9) | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  by Enzyme-linked immunosorbent assays; The values of intra- and inter-assay coefficients were around 5%. Concentration is expressed as ng/ml
plasma cell-free DNA by Real-time quantative PCR | Change from baseline, at after 6 weeks of HBOT and at after 6 times of neuropsychological treatment.
  DNA will be extracted from 200μL plasma samples with use of a QIAamp Blood Kit (Qiagen) according to the "blood and body fluid protocol" as recommended by the manufacturer. Plasma DNA will be measured by a real-time quantitative PCR assay for the β-globin gene and ND2 gene. The β-globin gene is present in all nucleated cells of the body while ND2 gene is specific mitochondrial DNA. Expression of β-globin and mtDNA will be measured by quantitative RT-PCR based on continuous measurements of Syber green fluorescent dye that binds to double stranded DNA generated during PCR and a specific primer pair for β-globin-354F (5'-GTG CAC CTG ACT CCT GAG GAG A-3') and β-globin-455R (5'-CCT TGA TAC CAA CCT GCC CAG-3') and ND2 (forward：5'-CAC AGA AGC TGC CAT CAA GTA -3'; reverse：5'-CCG GAG AGT ATA TTG TTG AAG AG -3').

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Tang Hsieh, MD, Study Chair — Chang Gung Medical Foundation
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We plan individual participant data sets to be shared while asking by other researchers.

REFERENCES:
- [Background] Maas AI, Stocchetti N, Bullock R. Moderate and severe traumatic brain injury in adults. Lancet Neurol. 2008 Aug;7(8):728-41. doi: 10.1016/S1474-4422(08)70164-9. PMID 18635021
- [Background] Lenzlinger PM, Morganti-Kossmann MC, Laurer HL, McIntosh TK. The duality of the inflammatory response to traumatic brain injury. Mol Neurobiol. 2001 Aug-Dec;24(1-3):169-81. doi: 10.1385/MN:24:1-3:169. PMID 11831551
- [Background] Zhang X, Chen Y, Jenkins LW, Kochanek PM, Clark RS. Bench-to-bedside review: Apoptosis/programmed cell death triggered by traumatic brain injury. Crit Care. 2005 Feb;9(1):66-75. doi: 10.1186/cc2950. Epub 2004 Sep 3. PMID 15693986
- [Background] Schmidt OI, Leinhase I, Hasenboehler E, Morgan SJ, Stahel PF. [The relevance of the inflammatory response in the injured brain]. Orthopade. 2007 Mar;36(3):248, 250-8. doi: 10.1007/s00132-007-1061-z. German. PMID 17333066
- [Background] Lu J, Goh SJ, Tng PY, Deng YY, Ling EA, Moochhala S. Systemic inflammatory response following acute traumatic brain injury. Front Biosci (Landmark Ed). 2009 Jan 1;14(10):3795-813. doi: 10.2741/3489. PMID 19273311
- [Background] Stein SC, Smith DH. Coagulopathy in traumatic brain injury. Neurocrit Care. 2004;1(4):479-88. doi: 10.1385/NCC:1:4:479. PMID 16174954
- [Background] Wang HC, Wang PM, Lin YJ, Kwan AL, Lin WC, Tsai NW, Cheng BC, Chang WN, Su BY, Kung CT, Lu CH. Serum adhesion molecules, outcome and neuro-psychological function in acute traumatic brain injury patients. Clin Chim Acta. 2013 Aug 23;423:122-9. doi: 10.1016/j.cca.2013.04.023. Epub 2013 Apr 30. PMID 23643853
- [Background] Lehnardt S. Innate immunity and neuroinflammation in the CNS: the role of microglia in Toll-like receptor-mediated neuronal injury. Glia. 2010 Feb;58(3):253-63. doi: 10.1002/glia.20928. PMID 19705460
- [Background] Rhind SG, Crnko NT, Baker AJ, Morrison LJ, Shek PN, Scarpelini S, Rizoli SB. Prehospital resuscitation with hypertonic saline-dextran modulates inflammatory, coagulation and endothelial activation marker profiles in severe traumatic brain injured patients. J Neuroinflammation. 2010 Jan 18;7:5. doi: 10.1186/1742-2094-7-5. PMID 20082712
- [Background] Carson MJ, Thrash JC, Walter B. The cellular response in neuroinflammation: The role of leukocytes, microglia and astrocytes in neuronal death and survival. Clin Neurosci Res. 2006 Dec;6(5):237-245. doi: 10.1016/j.cnr.2006.09.004. PMID 19169437
- [Background] Wang HC, Yang TM, Lin YJ, Chen WF, Ho JT, Lin YT, Kwan AL, Lu CH. Serial serum leukocyte apoptosis levels as predictors of outcome in acute traumatic brain injury. Biomed Res Int. 2014;2014:720870. doi: 10.1155/2014/720870. Epub 2014 Apr 17. PMID 24864256
- [Background] Kadhim HJ, Duchateau J, Sebire G. Cytokines and brain injury: invited review. J Intensive Care Med. 2008 Jul-Aug;23(4):236-49. doi: 10.1177/0885066608318458. Epub 2008 May 25. PMID 18504260
- [Background] Wang HC, Lin YJ, Shih FY, Chang HW, Su YJ, Cheng BC, Su CM, Tsai NW, Chang YT, Kwan AL, Lu CH. The Role of Serial Oxidative Stress Levels in Acute Traumatic Brain Injury and as Predictors of Outcome. World Neurosurg. 2016 Mar;87:463-70. doi: 10.1016/j.wneu.2015.10.010. Epub 2015 Oct 23. PMID 26481337
- [Background] Soriano SG, Piva S. Central nervous system inflammation. Eur J Anaesthesiol Suppl. 2008;42:154-9. doi: 10.1017/S0265021507003390. PMID 18289434
- [Background] Balabanov R, Goldman H, Murphy S, Pellizon G, Owen C, Rafols J, Dore-Duffy P. Endothelial cell activation following moderate traumatic brain injury. Neurol Res. 2001 Mar-Apr;23(2-3):175-82. doi: 10.1179/016164101101198514. PMID 11320596
- [Background] Wang HC, Lin YJ, Tsai NW, Su BY, Kung CT, Chen WF, Kwan AL, Lu CH. Serial plasma deoxyribonucleic acid levels as predictors of outcome in acute traumatic brain injury. J Neurotrauma. 2014 Jun 1;31(11):1039-45. doi: 10.1089/neu.2013.3070. Epub 2014 Mar 31. PMID 24467366
- [Background] Godman CA, Chheda KP, Hightower LE, Perdrizet G, Shin DG, Giardina C. Hyperbaric oxygen induces a cytoprotective and angiogenic response in human microvascular endothelial cells. Cell Stress Chaperones. 2010 Jul;15(4):431-42. doi: 10.1007/s12192-009-0159-0. Epub 2009 Dec 1. PMID 19949909
- [Background] Awasthi D, Church DF, Torbati D, Carey ME, Pryor WA. Oxidative stress following traumatic brain injury in rats. Surg Neurol. 1997 Jun;47(6):575-81; discussion 581-2. doi: 10.1016/s0090-3019(96)00461-2. PMID 9167783
- [Background] Tyurin VA, Tyurina YY, Borisenko GG, Sokolova TV, Ritov VB, Quinn PJ, Rose M, Kochanek P, Graham SH, Kagan VE. Oxidative stress following traumatic brain injury in rats: quantitation of biomarkers and detection of free radical intermediates. J Neurochem. 2000 Nov;75(5):2178-89. doi: 10.1046/j.1471-4159.2000.0752178.x. PMID 11032908
- [Background] Efrati S, Fishlev G, Bechor Y, Volkov O, Bergan J, Kliakhandler K, Kamiager I, Gal N, Friedman M, Ben-Jacob E, Golan H. Hyperbaric oxygen induces late neuroplasticity in post stroke patients--randomized, prospective trial. PLoS One. 2013;8(1):e53716. doi: 10.1371/journal.pone.0053716. Epub 2013 Jan 15. PMID 23335971
- [Background] Harch PG. Hyperbaric oxygen therapy for post-concussion syndrome: contradictory conclusions from a study mischaracterized as sham-controlled. J Neurotrauma. 2013 Dec 1;30(23):1995-9. doi: 10.1089/neu.2012.2799. Epub 2013 Oct 11. No abstract available. PMID 24004322
- [Background] Boussi-Gross R, Golan H, Fishlev G, Bechor Y, Volkov O, Bergan J, Friedman M, Hoofien D, Shlamkovitch N, Ben-Jacob E, Efrati S. Hyperbaric oxygen therapy can improve post concussion syndrome years after mild traumatic brain injury - randomized prospective trial. PLoS One. 2013 Nov 15;8(11):e79995. doi: 10.1371/journal.pone.0079995. eCollection 2013. PMID 24260334
- [Background] Chen CY, Wu RW, Tsai NW, Lee MS, Lin WC, Hsu MC, Huang CC, Lai YR, Kung CT, Wang HC, Su YJ, Su CM, Hsiao SY, Cheng BC, Chiang YF, Lu CH. Increased circulating endothelial progenitor cells and improved short-term outcomes in acute non-cardioembolic stroke after hyperbaric oxygen therapy. J Transl Med. 2018 Sep 12;16(1):255. doi: 10.1186/s12967-018-1629-x. PMID 30208940
- [Background] Kendall AC, Whatmore JL, Harries LW, Winyard PG, Eggleton P, Smerdon GR. Different oxygen treatment pressures alter inflammatory gene expression in human endothelial cells. Undersea Hyperb Med. 2013 Mar-Apr;40(2):115-23. PMID 23682543
- [Background] Chen Y, Nadi NS, Chavko M, Auker CR, McCarron RM. Microarray analysis of gene expression in rat cortical neurons exposed to hyperbaric air and oxygen. Neurochem Res. 2009 Jun;34(6):1047-56. doi: 10.1007/s11064-008-9873-8. Epub 2008 Nov 18. PMID 19015983
- [Background] Lin KC, Niu KC, Tsai KJ, Kuo JR, Wang LC, Chio CC, Chang CP. Attenuating inflammation but stimulating both angiogenesis and neurogenesis using hyperbaric oxygen in rats with traumatic brain injury. J Trauma Acute Care Surg. 2012 Mar;72(3):650-9. doi: 10.1097/TA.0b013e31823c575f. PMID 22491549
- [Background] Zhang JH, Lo T, Mychaskiw G, Colohan A. Mechanisms of hyperbaric oxygen and neuroprotection in stroke. Pathophysiology. 2005 Jul;12(1):63-77. doi: 10.1016/j.pathophys.2005.01.003. PMID 15869872
- [Background] Vlodavsky E, Palzur E, Soustiel JF. Hyperbaric oxygen therapy reduces neuroinflammation and expression of matrix metalloproteinase-9 in the rat model of traumatic brain injury. Neuropathol Appl Neurobiol. 2006 Feb;32(1):40-50. doi: 10.1111/j.1365-2990.2005.00698.x. PMID 16409552
- [Background] Huang L, Obenaus A. Hyperbaric oxygen therapy for traumatic brain injury. Med Gas Res. 2011 Sep 6;1(1):21. doi: 10.1186/2045-9912-1-21. PMID 22146562
- [Background] Chen Z, Ni P, Lin Y, Xiao H, Chen J, Qian G, Ye Y, Xu S, Wang J, Yang X. Visual pathway lesion and its development during hyperbaric oxygen treatment: a bold- fMRI and DTI study. J Magn Reson Imaging. 2010 May;31(5):1054-60. doi: 10.1002/jmri.22142. PMID 20432338
- [Background] May M, Milders M, Downey B, Whyte M, Higgins V, Wojcik Z, Amin S, O'Rourke S. Social Behavior and Impairments in Social Cognition Following Traumatic Brain Injury. J Int Neuropsychol Soc. 2017 May;23(5):400-411. doi: 10.1017/S1355617717000182. Epub 2017 Apr 12. PMID 28399953
- [Background] Milders M, Ietswaart M, Crawford JR, Currie D. Social behavior following traumatic brain injury and its association with emotion recognition, understanding of intentions, and cognitive flexibility. J Int Neuropsychol Soc. 2008 Mar;14(2):318-26. doi: 10.1017/S1355617708080351. PMID 18282329
- [Background] Allerdings MD, Alfano DP. Neuropsychological correlates of impaired emotion recognition following traumatic brain injury. Brain Cogn. 2006 Mar;60(2):193-4. doi: 10.1016/j.bandc.2004.09.018. PMID 16646115
- [Background] Tousignant B, Jackson PL, Massicotte E, Beauchamp MH, Achim AM, Vera-Estay E, Bedell G, Sirois K. Impact of traumatic brain injury on social cognition in adolescents and contribution of other higher order cognitive functions. Neuropsychol Rehabil. 2018 Apr;28(3):429-447. doi: 10.1080/09602011.2016.1158114. Epub 2016 Mar 10. PMID 26963905
- [Background] Sirois K, Tousignant B, Boucher N, Achim AM, Beauchamp MH, Bedell G, Massicotte E, Vera-Estay E, Jackson PL. The contribution of social cognition in predicting social participation following moderate and severe TBI in youth. Neuropsychol Rehabil. 2019 Oct;29(9):1383-1398. doi: 10.1080/09602011.2017.1413987. Epub 2017 Dec 18. PMID 29254438
- [Background] Westerhof-Evers HJ, Visser-Keizer AC, Fasotti L, Schonherr MC, Vink M, van der Naalt J, Spikman JM. Effectiveness of a Treatment for Impairments in Social Cognition and Emotion Regulation (T-ScEmo) After Traumatic Brain Injury: A Randomized Controlled Trial. J Head Trauma Rehabil. 2017 Sep/Oct;32(5):296-307. doi: 10.1097/HTR.0000000000000332. PMID 28786854
- [Background] Hart T, Brockway JA, Maiuro RD, Vaccaro M, Fann JR, Mellick D, Harrison-Felix C, Barber J, Temkin N. Anger Self-Management Training for Chronic Moderate to Severe Traumatic Brain Injury: Results of a Randomized Controlled Trial. J Head Trauma Rehabil. 2017 Sep/Oct;32(5):319-331. doi: 10.1097/HTR.0000000000000316. PMID 28520666
- [Background] Ali A, Hall I, Blickwedel J, Hassiotis A. Behavioural and cognitive-behavioural interventions for outwardly-directed aggressive behaviour in people with intellectual disabilities. Cochrane Database Syst Rev. 2015 Apr 7;2015(4):CD003406. doi: 10.1002/14651858.CD003406.pub4. PMID 25847633